CLINICAL TRIAL: NCT05867537
Title: Proof of Concept Human Study: Dietary Intervention to Modify Intestinal Inflammation in IBD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); Lithuanian University of Health Sciences (Other); University Medical Center Groningen, Netherland (Unknown); Weizmann Institute of Science, Israel (Unknown); Catholic University of the Sacred Heart (Other); Eurice European Research and project office GMBH, Germany (Unknown); Orebro University, Sweden (Unknown); Region Capital Denmark (Other); European Federation of Crohn´s and Ulcerative Colitis Associations, Belgium (Unknown)
Responsible Party: Principal Investigator, Samuel Huber, Director of the I. Department of Medicine, Prof. Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: miGut Health
Record Dates: First submitted 2023-04-03; First posted 2023-05-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Reduction of Intestinal Inflammatory Activity
Keywords: IBD; PSC
MeSH Terms: interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gluten-free diet in Crohn disease (Active Comparator)
  Interventions: Dietary Supplement: Gluten-free diet
- Gluten-free diet in ulcerative colitis (Active Comparator)
  Interventions: Dietary Supplement: Gluten-free diet
- Gluten-free diet in Primary sclerosing cholangitis (Active Comparator)
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — Implementation a 78-week dietary intervention to patients with ulcerative colitis, crohn´s disease and UC patients with associated PSC (PSC-IBD).

SUMMARY:
The objective of this clinical study is to demonstrate efficacy and feasibility of a long-term dietary intervention to modify intestinal inflammation in high-risk patient cohorts. To this end a 78 weeks wheat protein-free diet will be administered in patients with inflammatory bowel disease (IBD) with and without associated primary sclerosing cholangitis (PSC-IBD).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC, CD or PSC-IBD
* Willingness, to follow a gluten-free diet for 78 weeks
* Stable therapeutic treatment for more 8 weeks
* For CD: Harvey Bradshaw index (HBI) of more 5 points, corresponding to a minimum of mild intestinal inflammation in CD
* For UC: Mayo Score of more 2 points, corresponding to a minimum of mild intestinal inflammation in UC
* Patient signed informed consent

Exclusion Criteria:

* Antibiotics during last 4 weeks
* Intake of probiotics
* Gluten-free diet is already practiced
* Concomitant diagnosis of celiac disease
* Positive serology for transglutaminase IgA / IgG antibody or deamidated gliadin IgA / IgG
* Breast feeding
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical and endoscopic parameters of intestinal inflammation following 78 weeks of long-term gluten free dietary intervention, compared to pre-interventional levels in crohn´s disease (CD) | 78 Weeks + 12 Month follow-up
  Change of Harvey bradshaw index (HBI) for CD following 78 weeks of long-term gluten free dietary intervention. HBI range from 0 to 18 points + number of daily liquid stools (remission: HBI < 5, active disease: HBI ≥ 5, severe disease: HBI ≥ 8)
Change in clinical and endoscopic parameters of intestinal inflammation following 78 weeks of long-term gluten free dietary intervention, compared to pre-interventional levels in ulcerative colitis (UC) and PSC-IBD | 78 Weeks + 12 Month follow-up
  Change of partial Mayo Score (pMS) for UC and PSC-IBD following 78 weeks of long-term gluten free dietary intervention. pMS range from 0 to 12 points (remission: pMS < 2, mild activity: pMS 2-4, moderate activity: pMS 5-7, severe activity: pMS > 7).

SECONDARY OUTCOMES:
The efficacy and feasibility of a long-term dietary intervention to change mucosal transcripts of TNF-alpha of the intestine in IBD patients | 78 Weeks + 12 Month follow-up
  Changes between baseline and end of dietary period in TNF-alpha of mucosal transcript profiles.
The efficacy and feasibility of a long-term dietary intervention to change mucosal transcripts of IL-10 of the intestine in IBD patients | 78 Weeks + 12 Month follow-up
  Changes between baseline and end of dietary period in IL-10 mucosal transcript profiles.
The efficacy and feasibility of a long-term dietary intervention to change mucosal transcripts of IL-6 of the intestine in IBD patients | 78 Weeks + 12 Month follow-up
  Changes between baseline and end of dietary period in IL-6 mucosal transcript profiles.
Long-term dietary influence on intestinal microbiome in IBD patient cohorts | 78 Weeks + 12 Month follow-up
  Changes between baseline and end of dietary period in luminal microbiome dynamics from faecal samples identified by 16S RNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No